CLINICAL TRIAL: NCT05653687
Title: A Randomized, Monocentric Investigator-initiated Clinical Investigation Comparing Fluoroscopy Versus Freehand in Total Hip Arthroplasty
Brief Title: Total Hip Arthroplasty: Fluoroscopy vs Freehand
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ente Ospedaliero Cantonale, Bellinzona (Other)
Responsible Party: Principal Investigator, Christian Candrian, Principal Investigator, Ente Ospedaliero Cantonale, Bellinzona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORL-ORT-036
Record Dates: First submitted 2022-12-06; First posted 2022-12-16 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Intraoperative Fluoroscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fluoroscopy (Experimental)
  Interventions: Device: Intraoperative fluoroscopy
- Freehand (No Intervention)

INTERVENTIONS:
Device: Intraoperative fluoroscopy — Fluoroscopy is a medical procedure that makes a real-time video of the movements inside a part of the body by passing x-rays through the body over a period of time.
  Arms: Fluoroscopy

SUMMARY:
The aim of the study is to compare total hip arthroplasty intervention executed with or without the use of intraoperative fluoroscopy in terms of positioning of the hip prosthesis. The comparison will be made on post-operative follow-up X-ray performed as per clinical practice, in order to verify if intraoperative fluoroscopy provides better prosthesis components positioning or not.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing unilateral primary THA through DAA
* Patients aged 18-90 years old.
* Patients with a BMI >18 and <35.
* Patients able to provide informed consent.
* Informed consent as documented by signature.

Exclusion Criteria:

* Revision THA.
* Women who are pregnant or breast feeding.
* Presence of other clinically significant concomitant disease states (ASA IV).
* Previous enrolment into the current study.
* Enrolment of the investigator, his/her family members, employees and other dependent persons.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Acetabular component anteversion | 2 months post-operative
  Acetabular component anteversion will be measured on post-operative control antero-posterior pelvis view X-ray performed as per clinical practice using the PACS software according to the method described by Lewinnek et al. This method is based on the following equation to measure radiographic anteversion β.
  β = arcsin(S/L)
  Where S is the length of the short axis and L is the length of long axis of the ellipse. The ellipse is formed by the outer ring of the acetabulum component on the anteroposterior pelvis view X-ray.

CONTACTS AND LOCATIONS:
Locations (1):
- Ente Ospedaliero Cantonale, Lugano, Canton Ticino, Switzerland